CLINICAL TRIAL: NCT07051564
Title: A Clinical Study to Evaluate the Safety, Initial Efficacy and Pharmacokinetics of a Generic CNK-UT009 Cell Injection for the Treatment of Type 1 Diabetes Mellitus
Brief Title: Clinical Study on the Treatment of Type 1 Diabetes With CNK-UT009 Cell Injection
Acronym: CNK-UT009
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zibo Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.NO.070-1; GCP-250106-004 (Other: Zibo central hospital)
Record Dates: First submitted 2025-03-07; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 diabetes; CNK-UT009
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This is a single-arm, open, investigator-initiated clinical study of CNK-UT009 cell injection in pat (Experimental): This is a single-arm, open, investigator-initiated clinical study of CNK-UT009 cell injection in patients with type 1 diabetes. The purpose of this study is to evaluate the safety and tolerability of CNK-UT009 cell injection in patients with type 1 diabetes mellitus, determine the maximum tolerated dose (MTD), and evaluate the initial therapeutic effectiveness, PK characteristics and immunogenicity of CNK-UT009 cell injection. And the effect of CNK-UT009 cell injection on peripheral blood immune cells and serum cytokines.
  Interventions: Biological: CNK-UT009 cell injection

INTERVENTIONS:
Biological: CNK-UT009 cell injection — CNK-UT009 cell injection

SUMMARY:
This is a single-arm, open, investigator-initiated clinical study of CNK-UT009 cell injection in patients with type 1 diabetes. The purpose of this study is to evaluate the safety and tolerability of CNK-UT009 cell injection in patients with type 1 diabetes mellitus, determine the maximum tolerated dose (MTD), and evaluate the initial therapeutic effectiveness, PK characteristics and immunogenicity of CNK-UT009 cell injection. And the effect of CNK-UT009 cell injection on peripheral blood immune cells and serum cytokines.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of CNK-UT009 cell injection in the treatment of patients with type 1 diabetes and to determine the maximum tolerated dose (MTD).

Secondary objectives include:

1. Assessing the preliminary efficacy of CNK-UT009 cell injection in treating patients with type 1 diabetes;
2. Evaluating the pharmacokinetic (PK) characteristics of CNK-UT009 cell injection;
3. Assessing the impact of CNK-UT009 cell injection reinfusion on peripheral blood immune cells;
4. Assessing the impact of CNK-UT009 cell injection reinfusion on serum cytokines;
5. Evaluating the immunogenicity of CNK-UT009 cell injection.

The primary endpoints of this clinical trial are:

1. Safety and tolerability endpoints: Adverse events occurring after the reinfusion of CNK-UT009 cell injection, including the type, frequency, and severity of treatment-emergent adverse events (TEAEs), to determine the maximum dose-limiting toxicity (DLT) and tolerated dose (MTD);
2. Primary efficacy endpoint: Changes in serum C-peptide peak and area under the curve (AUC) after a 2-hour mixed meal tolerance test (MMTT) before and after the reinfusion of CNK-UT009 cell injection.

Secondary research endpoints are:

1. Secondary efficacy endpoints: Changes in the percentage of glycated hemoglobin (HbA1c) before and after the reinfusion of CNK-UT009 cell injection;
2. Before and after the reinfusion of CNK-UT009 cell injection, the patient wore a continuous glucose monitoring system (CGM), measuring average glucose levels, time in range (TIR), time above range (TAR), and changes in time below range (TBR);
3. Changes in the average daily insulin dosage within 7 days before and after the reinfusion of CNK-UT009 cell injection;
4. Changes in the titer of islet autoantibodies before and after the reinfusion of CNK-UT009 cell injection.

Pharmacokinetics (PK): Changes in the number of CAR-positive cells in peripheral blood before and after the reinfusion of CNK-UT009 cell injection, and the dynamic changes in DNA copy number of T cells.

Peripheral blood immune cells: Subtypes of immune cells in peripheral blood before and after the reinfusion of CNK-UT009 cell injection, including but not limited to NKG2D-L (MICA/B, ULBP1/2/3/5/6) + T cells, B cells, and changes in the percentage of Treg cells.

Serum cytokines: Changes in serum cytokines (including IL2) before and after the reinfusion of CNK-UT009 cell injection, including IL6, IL10, IFN-γ, TNF-α, etc.

Immunogenicity: The binding ratio of CNK-UT009 cell injection to serum antibodies (IgG) in the subjects and the rate of change.

ELIGIBILITY:
Inclusion criteria

Patients who meet all of the following criteria can be considered for inclusion:

* Age 18 to 65 years old (including the cut-off value), gender not limited;
* Diagnosed with autoimmune type 1 diabetes (meeting the diagnostic criteria of the "Chinese Guidelines for the Diagnosis and Treatment of Type 1 Diabetes (2021 Edition)"), and the peak C-peptide was ≥0.2nmol/L after 2-hour mixed meal (MMTT) stimulation during the screening period;
* At least one insulin autoantibody is positive, such as glutamate decarboxylase autoantibody (GADA), protein tyrosine phosphatase autoantibody (IA-2A), insulin autoantibody (IAA) (without insulin use or within 2 weeks of insulin treatment), zinc transporter antibody (ZnT8A);
* Glycated hemoglobin (HbA1c) ≥6.5% and ≤10.5%;
* Body mass Index (BMI)≥18kg/m ² and ≤35kg/m ²;
* Have sufficient organ and bone marrow functions, and the laboratory test values within 7 days before enrollment meet the following requirements, as detailed below:

Blood routine: Absolute neutrophil count (ANC) ≥1.0× 109 /L; Absolute lymphocyte count (LYC) ≥1.0× 109 /L; Platelet count (PLT) ≥75×109/L; Hemoglobin content (HGB) ≥80g/L; Heart: Left ventricular ejection fraction (LVEF) ≥50%; Cardiac function grade 1-2 Lung function: Indoor blood oxygen saturation ≥92%; Liver function: Serum total bilirubin (TBIL) ≤1.5×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN; Renal function: Serum creatinine (Cr) ≤1.5×ULN; Glomerular filtration rate (eGFR) ≥60mL/min/1.73m2 (calculated by the MDRD formula)

* For female patients of childbearing age, the serum or urine pregnancy result must be negative before enrollment, and they must agree to take acceptable measures to minimize the possibility of pregnancy during the trial. Female patients of childbearing age or male patients whose sexual partners are female patients of childbearing age need to take effective contraceptive measures throughout the treatment period and 6 months after the last medication.
* Agree to abide by the principles and suggestions of medical nutrition therapy in the "Chinese Guidelines for the Diagnosis and Treatment of Type 1 Diabetes Mellitus (2021 Edition)";
* Voluntarily participate in clinical research, understand and be informed of this study, sign the informed consent form, and be willing to follow all trial procedures.

Exclusion criteria

Patients meeting any of the following criteria are not eligible for enrollment:

* Active malignant tumors requiring treatment, except for non-melanoma skin cancer or carcinoma in situ (such as breast, cervical);
* Subjects who have received organ transplants in the past or are preparing to receive organ transplants;
* Those who have received immunosuppressant treatment within 4 weeks before enrollment and/or require long-term immunosuppressive treatment during the study period, and are allowed to use topical, inhaled or intranasal corticosteroids intermittently;
* Any life-threatening bleeding events occurred within 3 months before enrollment, including the need for blood transfusion treatment, surgery or local treatment, and continuous drug treatment;
* A history of arterial or venous thromboembolic events within 6 months before enrollment, including myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other serious thromboembolic events. Thrombosis derived from implantable venous infusion ports or catheters, or superficial venous thrombosis, is excluded if the thrombus is stable after conventional anticoagulant therapy. Prophylactic use of small doses of low-molecular-weight heparin (such as enoxaparin 40 mg/ day) is permitted;
* Severe bleeding tendency or coagulation dysfunction, or currently undergoing thrombolytic therapy;
* Uncontrollable hypertension, with a systolic blood pressure greater than 160 mmHg or a diastolic blood pressure greater than 100 after the best medical treatment mmHg, history of hypertensive crisis or hypertensive encephalopathy;
* Symptomatic congestive heart failure (New York Heart Association Classification II-IV). Symptomatic or poorly controlled arrhythmias. A history of congenital long QT syndrome or corrected QTc>500 ms during screening;
* Pulmonary diseases such as a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, and severe impairment of lung function;
* Active pulmonary tuberculosis (TB), those who are currently undergoing anti-tuberculosis treatment or have received anti-tuberculosis treatment within one year prior to the first administration of medication; Active hepatitis B and C virus carriers, human immunodeficiency virus carriers, and known syphilis carriers;
* There was a severe infection in the active stage or with poor clinical control within 4 weeks before enrollment, including but not limited to hospitalization due to infection, bacteremia or severe pneumonia complications;
* Complications of diabetes, such as:

  1. Ketoacidosis
  2. Renal insufficiency (urine protein ≥2+, eGFR<60mL/min/1.73m2);
  3. Active or untreated proliferative retinopathy;
  4. Diabetic foot ulcer
  5. Amputation caused by diabetes;
  6. Severe peripheral neuropathy.
* Have received any non-insulin hypoglycemic drugs or drugs that affect glucose metabolism within 4 weeks or 5 half-lives (of the drug) before enrollment, whichever is shorter.
* Two or more severe and unexplained hypoglycemic events occurred within 6 months before enrollment;
* A history of inability to complete the mixed meal tolerance test (MMTT), or a significant allergic reaction (such as anaphylactic shock) to any component in the mixed meal of the MMTT test;
* Received treatment from other clinical studies within 4 weeks before enrollment;
* Those who have received attenuated live vaccines within 4 weeks before enrollment;
* Those who have used any gene therapy products in the past;
* It is known to be allergic to any component of CNK-UT009 cell injection;
* Suffering from a known mental illness or substance abuse disorder, and these disorders may interfere with the subject's ability to cooperate with the research requirements;
* Subjects whose researchers consider to have other life-threatening serious complications that may potentially or interfere with the assessment of this study;
* Other circumstances that the researcher deems inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CNK-UT009 cell injection for the treatment of patients with type 1 diabetes Evaluation of the safety and tolerability of the user | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  Safety and tolerability endpoints: Adverse events that occurred after reinfusion of CNK-UT009 cell injection. The type, occurrence frequency and severity of (TEAE) determine that dose-limiting toxicity (DLT) is the greatest Tolerated dose (MTD)
CNK-UT009 cell injection for the treatment of patients with type 1 diabetes Evaluation of the effectiveness of it | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  The primary efficacy endpoint: A 2-hour mixed meal tolerance test before and after reinfusion of CNK-UT009 cell injection The changes of the peak value of serum C-peptide and the area under the curve (AUC) after stimulation by (MMTT)

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) characteristics of CNK-UT009 cell injection | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  peak concentration (Cmax)
To evaluate the pharmacokinetic (PK) characteristics of CNK-UT009 cell injection | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  half-life (T1/2)
To evaluate the pharmacokinetic (PK) characteristics of CNK-UT009 cell injection | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  Time to peak (Tmax)
To evaluate the pharmacokinetic (PK) characteristics of CNK-UT009 cell injection | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  systemic clearance rate (CL)
To evaluate the pharmacokinetic (PK) characteristics of CNK-UT009 cell injection | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  Volume of distribution (Vd)
To evaluate the pharmacokinetic (PK) characteristics of CNK-UT009 cell injection | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  Area under the blood drug concentration-time curve (AUC）
CNK-UT009 cell injection for the treatment of patients with type 1 diabetes Evaluation of peripheral blood immune cell subsets of the patient | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  The changes in the percentages of immune cell subsets in peripheral blood before and after the reinfusion of CNK-UT009, including but not limited to NKG2D-L(MICA/B, ULBP1/2/3/5/6) +T cells, B cells, Treg cells
CNK-UT009 cell injection for the treatment of patients with type 1 diabetes Evaluation of serum cytokines of the patient | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  The changes of serum cytokines before and after reinfusion of CNK-UT009, including IL2, IL6, IL10, IFN-γ, and TNF-α Wait.
CNK-UT009 cell injection for the treatment of patients with type 1 diabetes Evaluation of the immunogenicity of the individual | The first cycle lasts for 21 days. The second to the fourth cycles each last for 14 days. The treatment follow-up period lasted for a total of 12 months
  The binding ratio of antibodies (IgG) between CNK-UT009 cell injection and the serum of the subjects is directly reflected. The changes of antibody-mediated rejection (AMR) of the test subjects to the CNK-UT009 cell injection.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Pang, Doctor, Principal Investigator — Zibo Central Hospital
Locations (1):
- Zibo Central hospital, Zibo, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
We will disclose the safety and tolerability data of CNK-UT009 cell injection in the treatment of patients with type 1 diabetes, and elaborate on the maximum tolerated dose (MTD), the initial therapeutic effect, PK characteristics and immunogenicity of CNK-UT009 cell injection, as well as its impact on peripheral blood immune cells and serum cytokines.
Supporting Information: SAP, Analytic Code
Time Frame: December 2025 -December 2027
Access Criteria: We will make our IPD data public by publishing academic papers. Everyone can download the articles from the official websites of relevant journals to obtain our data。